CLINICAL TRIAL: NCT03551717
Title: Retinal Microvascularization and Cardiovascular Diseases
Brief Title: Retinal Microvascularization and Cardiovascular Disease
Acronym: NESTOR
Status: Terminated | Type: Observational
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MEILLON AOI 2017
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: High Cardiovascular Risk Patients; Low Cardiovascular Risk Patients
MeSH Terms: interventions — Optical Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High cardiovascular risk patients: Adult patients hospitalized in the Cardiology Department of the University Hospital of Dijon Burgundy for acute coronary syndrome, patients between D1 and D5 of acute coronary syndrome, who can be moved for an ophthalmology consultation where the retinal imaging is done (heart monitoring in the presence of an experienced cardiologist if necessary)
  Interventions: Other: Optical Coherence Tomography angiography; Other: Fundus; Other: cardiac ultrasound scan
- Low cardiovascular risk patients: Adult patients recruited in the Ophthalmology Department of the University Hospital of Dijon Burgundy following a standard consultation for cataract surgery.
  The age balance of the patients included in the two groups will be checked regularly.
  Interventions: Other: Optical Coherence Tomography angiography; Other: Fundus

INTERVENTIONS:
Other: Optical Coherence Tomography angiography — At the inclusion visit for all patients and at M3 only for 50 patients.
Other: Fundus — At the inclusion visit for all patients and at M3 only for 50 patients.
Other: cardiac ultrasound scan — Only for 50 patients, 3 months after the initial cardiovascular event
  Groups: High cardiovascular risk patients

SUMMARY:
The main objective of this study is to investigate whether there are links between the blood vessels of the retina as a whole and heart and/or vascular diseases (cardiovascular diseases).

The arteries and veins of the retina are, like the large vessels of the human body (aorta, coronary, cerebral arteries), exposed to the complications of hypertension, diabetes, obesity, dyslipidemia (abnormal blood lipid profile) or tobacco. Several studies have shown that changes in retinal vessels (microvascularization) generally occur several years before damage to large peripheral vessels (macrovascularization). The study of the vessels of the retina is now possible thanks to simple and non-invasive examinations of photographs (not creating any lesion). They allow a painless evaluation of the vessels in the retina.

Ultimately, if this study is conclusive, the patient's cardiovascular risk could be evaluated simply by analysis of the vessels of the retina.

The study is being conducted in the ophthalmology and cardiology departments of Dijon University Hospital. In total, the investigators wish to include approximately 510 patients who present cardiovascular risk factors (255 low risk patients recruited in the ophthalmology department and 255 high risk patients hospitalized in the cardiology department).

All patients participating in the study will be asked to visit the ophthalmology department for a complete examination of the retina.

ELIGIBILITY:
Inclusion Criteria:

* Person who gave oral consent
* High cardiovascular risk group: Adult patients hospitalized in the Cardiology Department of the University Hospital of Dijon Burgundy for acute coronary syndrome, patients between D1 and D5 of acute coronary syndrome, who can be moved for an ophthalmology consultation where the retinal imaging is done (heart monitoring in the presence of an experienced cardiologist if necessary)
* Low cardiovascular risk group: Adult patients over 40 years of age recruited in the Ophthalmology Department of the University Hospital of Dijon Burgundy following a standard consultation for cataract surgery, ocular surface pathologies and optical correction.

Exclusion Criteria:

* Person not affiliated to national health insurance
* Patient refusal
* Minor patient
* Protected patient
* Ophthalmological history (macular vascular or degenerative disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High and low cardiovascular risk patients
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Surface of the avascular zone in the central retina | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France